CLINICAL TRIAL: NCT05416424
Title: Effects of Implementing a Post-surgical Dietary and Lifestyle Protocol on Uterine Fibroid Recurrence
Brief Title: Life Study: Lifestyle Intervention in Fibroid Elimination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-00226
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Healthy patients aged 18-50 who have a uterus, identify as female and have come to the outpatient Center for Women's Health (CWH) for management of bleeding, pelvic pain and fibroids. They will be offered enrollment post-surgery or procedure and will be followed longitudinally for 12 months.
  Interventions: Other: LIFE program

INTERVENTIONS:
Other: LIFE program — During the nutritionist visits, subjects will be asked to discuss and evaluate their current diet and will be given recommended dietary changes. The recommended dietary changes include focusing on eating nutrient dense foods, staying consistent with the timing of meals, limiting added sugars, aiming to have balanced meals and snacks, being a mindful eater, and aiming to drink approximately 2 liters of water a day. Additionally, they will review the nutrition survey with the registered dietician. During the office visits with a doctor, subjects will be given exercise counseling. They will be asked to do 150 minutes per week of moderate intensity aerobic activity

SUMMARY:
The study will evaluate a lifestyle, nutrition, and exercise program to assess whether this program is acceptable and feasible for patients..Researchers will examine if the LIFE program can modify fibroid recurrence.

DETAILED DESCRIPTION:
This prospective cohort pilot study will enroll asymptomatic, post-surgical patients who underwent a laparoscopic, open, robotic myomectomy, or other procedure ie Sonata, Accessa for fibroid removal. Patients will be offered enrollment into a lifestyle, nutrition, supplement, and exercise program to assess whether this program is acceptable and feasible for patients. Surveys will be collected at 3-6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 18-50, who are seeking care at the Center for Fibroid Care at NYU
* Participants who have had a procedure or surgery performed to removed fibroids within the last 3 months and are now considered "fibroid free."
* Be English speaking and be able to read/write in English
* Visit with PCP within the last 3 months with labs

Exclusion Criteria:

* Currently Pregnant
* Use of any medication, hormonal or GNRH agonists, that would affect fibroid growth
* Postmenopausal women
* Non-English speaking
* Fibroid procedure or surgery outside of the 3-month window
* Women who are physically incapable of following a physical activity regimen
* Women with multiple dietary restrictions that would impact their ability to follow recommended dietary plan. (ie. GI disorders)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of LIFE program as measured by Self report survey | 12 month visit.
  Patient satisfaction survey will assess if patients found the program acceptable on a 5 point Likert scale ( not at all acceptable, fair, moderate, good excellent).
Change in improvement in quality of life as measured by Quality of Life Scale (QOLS) | Baseline, 6 month, 12 month
  The Quality of Life Scale (QOLS) was originally a 15-item instrument that measured five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation. Using a 7-point response scale, scores are summed so that a higher score indicates higher quality of life. The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112.
Change in fibroid recurrence as measured by standard of care ultrasounds | Baseline, 6 month, 12 month
  Adherence to a lifestyle program changes rate of fibroid recurrence as assessed by standard of care pelvic ultrasound results.

CONTACTS AND LOCATIONS:
Overall Officials: Taraneh Shirazian, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Taraneh.shirazian@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.